CLINICAL TRIAL: NCT00805103
Title: Hypofractionated Stereotactic Radiotherapy (HF-SRT) for Large-Volume Brain Metastases
Brief Title: Perfexion Brain Metastasis
Acronym: HF-SRT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 08-0602-C
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Brain Metastases
Keywords: Brain Metastases; Stereotactic radiosurgery (SRS); Hypofractionated stereotactic radiotherapy (HSRT); Recurrent Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- (HFA-SRT) in Large-Volume Brain Metastases (Experimental)
  Interventions: Radiation: Hypofractionated stereotactic radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated stereotactic radiotherapy — Patients will be initially administered 8 Gy RT (level). The dose at each level will be increase by 2 Gy up to level 4. If ≥ 2 of the patients in a dose cohort encounter a DLT, then that dose level will be declared the maximum administered dose. An additional 3 patients will then be entered at the previous dose level and provided no more than one patient experiences a DLT, that level will be declared the maximum tolerated dose (MTD). Up to 6 more patients can be treated at the given dose level while awaiting the results of 6 months of follow-up.

SUMMARY:
Brain metastases occur in 20% to 40% of all patients with cancer , with an incidence 10 times higher than that of primary malignant brain tumors. Patients with brain metastases have a poor prognosis with a median survival of 1-2 months with corticosteroids and 5-7 months with whole brain radiotherapy (WBRT). Local control achieved with WBRT in patients with otherwise controlled systemic disease remains at issue. A single high dose of radiation delivered with high precision to the target lesion (Stereotactic radiosurgery (SRS)), is considered standard care in salvage of recurrent lesions after WBRT. SRS can destroy tumour with very little damage to surrounding tissue. Research suggests that delivering radiotherapy in a number of smaller doses is more beneficial than receiving all of the radiotherapy in a single dose. Brain metastases are well suited for SRS as they are often small, radiographically well-circumscribed, pseudospherical tumors that are noninfiltrative.

DETAILED DESCRIPTION:
With increasing volume of tumor, the dose of radiosurgery that can be safely delivered to recurrent oligo-metastases in the brain must be reduced. However, reducing the dose of radiosurgery also compromises local control. There is mounting evidence of a local control benefit to a hypofractionated approach in radiation delivery for brain metastases compared with single fraction radiosurgery. Here we propose a novel therapeutic strategy that builds on this concept whereby time between each delivered fraction will enable us to measure and adapt to response, with the objective of reducing irradiated volumes and improving outcomes. In general, the treatment of malignant tumors benefits from fractionation of the dose due to a number of radiobiological properties (redistribution, reoxygenation, repair) that distinguish, and select against, malignant lesions in the fractionation process. Hypofractionated stereotactic radiotherapy (HSRT) is a method of delivering a highly conformal dose distribution in a few treatment sessions using a relocatable stereotactic frame. HSRT may be an attractive alternative to SRS because it may 1) improve patient comfort by removing the invasive nature of SRS frames, 2) confer a radiobiologic advantage over single fraction treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1-5 recurrent brain metastases after WBRT, and
* At least 1 lesions >2cm in maximum diameter
* ECOG 0-2
* Life expectancy >3months
* Age ≥ 18 years old

Exclusion Criteria:

* Edentulous patients
* Prior surgery or injury to hard palate
* Severe claustrophobia
* Contraindication to MRI
* Contraindication to IV contrast (Gadolinium) administration
* Other medical conditions that would preclude study investigations
* Prior radiosurgery to recurrent lesions
* Radiation cannot be delivered at the assigned dose level in a manner that respects OAR constraints (3.2.2.4.2.3.4) (e.g. lesions within brainstem or abutting optic structures)
* Any lesion >5cm in diameter, or total volume of tumor > 60cc
* Pregnant Women
* Men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
This study aims to determine what the maximum tolerated dose of hypofractionated adaptive stereotactic radiotherapy (HFA-SRT) for recurrent brain metastases is. | every 3 months for 3 years

SECONDARY OUTCOMES:
The secondary outcome will be to evaluate the overall survival and change in tumour response. | every 3 months for 3 years
Measure acute and late toxicities | every 3 months for 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Chung, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Toronto, Ontario, Canada